CLINICAL TRIAL: NCT04052308
Title: Decrease in Blood Pressure in PARQVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, Full Professor in Orthopedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPPesq 04019418700000068
Record Dates: First submitted 2019-08-02; First posted 2019-08-09 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis; Blood Pressure
Keywords: Knee Osteoarthritis; Blood Pressure; HIIT
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Two days of lectures about knee OA, but will also come to the hospital after the first class to consult about nutritional habits to be improved; therapy session with the psychologists, sessions with the physical therapy team; sessions with the physical educators team.
  They will be submitted to 24-hour ambulatory blood pressure monitoring (ABPM) at baseline and at the end fo the study; The arterial stiffness and endothelial reactivity will be assessed by measurement of the carotid-femoral pulse wave velocity by means of a non-invasive automatic device at baseline and at the end fo the study; Answer EQ-5D-5L at baseline and at the end fo the study.
  Interventions: Behavioral: ABPM; Behavioral: The arterial stiffness and endothelial reactivity; Behavioral: Euroqol EQ-5D-5L; Behavioral: Lectures about knee OA
- Continuous group (Experimental): Two days of lectures about knee OA, but will also come to the hospital after the first class to consult about nutritional habits to be improved; therapy session with the psychologists, sessions with the physical therapy team; sessions with the physical educators team. The supervised exercise sessions will consist of 10 min of warm-up stretching exercises, 40 min of treadmill (40 min on treadmill at 60% of reserve heart rate), 20 min of sub-maximal strength training and 10 min of cooling exercises. They will be submitted to 24-hour ambulatory blood pressure monitoring (ABPM) at baseline and at the end of the study. The arterial stiffness and endothelial reactivity will be assessed by measurement of the carotid-femoral pulse wave velocity by means of a non-invasive automatic device at baseline and at the end of the study.
  Interventions: Behavioral: ABPM; Behavioral: The arterial stiffness and endothelial reactivity; Behavioral: Euroqol EQ-5D-5L; Behavioral: Lectures about knee OA; Behavioral: Continuous intensity exercise
- Interval group (Experimental): Two days of lectures about knee OA, but will also come to the hospital after the first class to consult about nutritional habits to be improved; therapy session with the psychologists, sessions with the physical therapy team; sessions with the physical educators team. The supervised exercise sessions will consist of 10 min of warm-up stretching exercises, 40 min of treadmill (40 min on treadmill with alternating intensity between 50% and 80%) of HR, resulting in an average load of 60% ((50% 2) + 80% 3)), 20 min of sub-maximal strength training and 10 min of cooling exercises. They will be submitted to 24-hour ambulatory blood pressure monitoring (ABPM) at baseline and at the end of the study. The arterial stiffness and endothelial reactivity will be assessed by measurement of the carotid-femoral pulse wave velocity by means of a non-invasive automatic device at baseline and at the end of the study.
  Interventions: Behavioral: ABPM; Behavioral: The arterial stiffness and endothelial reactivity; Behavioral: Euroqol EQ-5D-5L; Behavioral: Lectures about knee OA; Behavioral: Exercises with varying intensity and interval

INTERVENTIONS:
Behavioral: ABPM — Ambulatory Blood Pressure Monitoring at Baseline and at the end of the study
Behavioral: The arterial stiffness and endothelial reactivity — The arterial stiffness and endothelial reactivity will be assessed at baseline and at the end of the study
Behavioral: Euroqol EQ-5D-5L — Answer Euroqol EQ-5D-5L at baseline and at the end of the study
Behavioral: Lectures about knee OA — Patients will participate in two days of lectures two-months apart on the subject of knee OA, but will also come to the hospital at months 1, 3 and 5 after the first class to consult about nutritional habits to be improved; at months 4 and 6 to participate in a group therapy session with the psychologists, 7 sessions with the physical therapy team followed by 7 sessions with the physical educators team (once a week/4 weeks and once every two weeks, three times).
Behavioral: Continuous intensity exercise — 40 min of treadmill physical exercise (40 min on treadmill at 60% of reserve heart rate.)
  Arms: Continuous group
Behavioral: Exercises with varying intensity and interval — 40 min of treadmill physical exercise ( 40 min on treadmill with alternating intensity between 50% (2 min) and 80% (1 min) of HR, resulting in an average load of 60% ((50% 2) + 80% / 3)), 20 min of sub-maximal strength training and 10 min of cooling exercises.
  Arms: Interval group

SUMMARY:
The tripod of OA clinical treatment is education, weight loss and exercise. A sedentary lifestyle has been characterized as an independent risk factor for cardiovascular disease. Studies have shown the inverse association between the level of physical activity and the incidence of cardiovascular disease. High Intensity Interval Training (HIIT), which consists of repeated high-intensity exercise sessions interspersed with passive recovery. Active, has been studied as a new therapeutic approach and has been shown to be effective in controlling blood pressure (BP) and arterial stiffness in treated hypertensive individuals. HIIT training has also been shown to be able to reverse the hemodynamic, metabolic and hormonal changes that are involved in the pathophysiology of essential hypertension, leading to improved arterial stiffness and BP response, endothelin-1 and nitrite / nitrate to exercise, increased cardiorespiratory fitness when compared to moderate-intensity continuous exercise in young women with a family history of essential hypertension. Six weeks of HIIT training (3 times / week) reduced body fat and waist circumference in young women. , while increasing fat-free mass, maximum running speed and aerobic fitness. Two recent studies evaluating body weight change in overweight patients have shown that HIIT training is comparable to moderate-intensity continuous exercise, but HIIT is more efficient compared to time spent training, which may facilitate the inclusion of daily routine training of patients. Previous work performed by the authors patients undergoing an education and physical activity program showed improvement in WOMAC. The investigators believe that the inclusion of an HIIT training protocol may lead to improved BP and hemodynamic variables in patients with knee osteoarthritis. To evaluate the effect of high intensity interval physical training associated with an educational program on BP, hemodynamic variables of individuals undergoing treatment for knee OA. 63 patients with knee OA will be randomized into 3 groups: interval exercise (21), continuous exercise (21) and control (21). Patients will be evaluated for BP using ABPM, arterial stiffness and endothelial reactivity by measuring carotid-femoral pulse wave velocity and quality of life using the Euroqol scale.

DETAILED DESCRIPTION:
High Intensity Interval Training (HIIT), which consists of repeated high intensity exercise sessions interspersed with passive / active recovery, has been studied as a new approach to hypertension therapy and systemic arterial hypertension. HIIT training has also been shown to be able to reverse how the hemodynamic, metabolic and hormonal changes that are involved in the physiology of essential hypertension, leading to improved arterial stiffness and BP response, endothelin-1 and nitrite / nitrate to exercise, Increased cardiorespiratory capacity when moderate-intensity continuous exercise was performed in young women with a history of essential arterial hypertension.

Six weeks of HIIT training (3 times / week) reduced body fat and waist circumference in young women while increasing fat-free mass, maximum running speed, and aerobic fitness. Two recent studies evaluating body constitution change in overweight patients have shown that HIIT training is comparable to moderate-intensity continuous exercise, but HIIT is more efficient compared to the time spent during training, and HIIT can deliver savings of approximately 40% of the training time, which can facilitate the inclusion of training in the daily routine of patients.

In previous work by the investigators, patients undergoing an education and physical activity program showed improvement in WOMAC. Researchers believe that the inclusion of an HIIT training protocol may lead to improved BP and hemodynamic variables in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with OAJ and SAH using antihypertensive medications
* Classified as Kelgreen and Lawrence grades I to III (K-L), ie any degree of gonarthritis without obliteration of the joint space.
* Indication of clinical treatment of OA.
* Patients not submitted to previous lower limb arthroplasty.
* Patients not submitted to knee infiltration up to 6 months before study.
* Patients without personal history of cognitive, psychiatric and / or neurological disorders, whose symptoms presented at the time of the evaluation are related or significantly interfere with the functions of attention, memory, logical reasoning, understanding, in order to impair the assimilation of the given guidelines.
* Patients who have not been doing regular physical activity (more than once a week) for the past 6 months.
* Patients able to perform physical activity from a cardiological point of view
* Ability to read, understand and answer the questionnaires.

Exclusion Criteria:

- Missing interventions and not performing the tasks determined by professionals.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Effects of high intensity exercise on blood pressure in individuals undergoing treatment for knee osteoarthritis | 16 weeks
  To assess the effect of high intensity versus continuous interval training of moderate intensity associated with an educational program on resting blood pressure.

SECONDARY OUTCOMES:
Effects of high intensity exercise on quality of life | 16 weeks
  Evaluate whether the high-intensity interval training associated with an educational program improves the quality of life evaluated through the Euroqol (ranging from 0 to 1, with higher score indicating better)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Ocampos, MD, Principal Investigator — University of São Paulo General Hospital

REFERENCES:
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Rillo O, Riera H, Acosta C, Liendo V, Bolanos J, Monterola L, Nieto E, Arape R, Franco LM, Vera M, Papasidero S, Espinosa R, Esquivel JA, Souto R, Rossi C, Molina JF, Salas J, Ballesteros F, Radrigan F, Guibert M, Reyes G, Chico A, Camacho W, Urioste L, Garcia A, Iraheta I, Gutierrez CE, Aragon R, Duarte M, Gonzalez M, Castaneda O, Angulo J, Coimbra I, Munoz-Louis R, Saenz R, Vallejo C, Briceno J, Acuna RP, De Leon A, Reginato AM, Moller I, Caballero CV, Quintero M. PANLAR Consensus Recommendations for the Management in Osteoarthritis of Hand, Hip, and Knee. J Clin Rheumatol. 2016 Oct;22(7):345-54. doi: 10.1097/RHU.0000000000000449. PMID 27660931
- [Background] Physical activity and cardiovascular health. NIH Consensus Development Panel on Physical Activity and Cardiovascular Health. JAMA. 1996 Jul 17;276(3):241-6. PMID 8667571
- [Background] Tanaka H, Dinenno FA, Monahan KD, Clevenger CM, DeSouza CA, Seals DR. Aging, habitual exercise, and dynamic arterial compliance. Circulation. 2000 Sep 12;102(11):1270-5. doi: 10.1161/01.cir.102.11.1270. PMID 10982542
- [Background] Cameron JD, Dart AM. Exercise training increases total systemic arterial compliance in humans. Am J Physiol. 1994 Feb;266(2 Pt 2):H693-701. doi: 10.1152/ajpheart.1994.266.2.H693. PMID 8141370
- [Background] Kakiyama T, Sugawara J, Murakami H, Maeda S, Kuno S, Matsuda M. Effects of short-term endurance training on aortic distensibility in young males. Med Sci Sports Exerc. 2005 Feb;37(2):267-71. doi: 10.1249/01.mss.0000152733.12578.5a. PMID 15692323
- [Background] Guimaraes GV, Ciolac EG, Carvalho VO, D'Avila VM, Bortolotto LA, Bocchi EA. Effects of continuous vs. interval exercise training on blood pressure and arterial stiffness in treated hypertension. Hypertens Res. 2010 Jun;33(6):627-32. doi: 10.1038/hr.2010.42. Epub 2010 Apr 9. PMID 20379194
- [Background] Ciolac EG, Bocchi EA, Bortolotto LA, Carvalho VO, Greve JM, Guimaraes GV. Effects of high-intensity aerobic interval training vs. moderate exercise on hemodynamic, metabolic and neuro-humoral abnormalities of young normotensive women at high familial risk for hypertension. Hypertens Res. 2010 Aug;33(8):836-43. doi: 10.1038/hr.2010.72. Epub 2010 May 7. PMID 20448634
- [Background] Hazell TJ, Hamilton CD, Olver TD, Lemon PW. Running sprint interval training induces fat loss in women. Appl Physiol Nutr Metab. 2014 Aug;39(8):944-50. doi: 10.1139/apnm-2013-0503. Epub 2014 Mar 18. PMID 24905559
- [Background] Wewege M, van den Berg R, Ward RE, Keech A. The effects of high-intensity interval training vs. moderate-intensity continuous training on body composition in overweight and obese adults: a systematic review and meta-analysis. Obes Rev. 2017 Jun;18(6):635-646. doi: 10.1111/obr.12532. Epub 2017 Apr 11. PMID 28401638
- [Background] Zhang H, Tong TK, Qiu W, Zhang X, Zhou S, Liu Y, He Y. Comparable Effects of High-Intensity Interval Training and Prolonged Continuous Exercise Training on Abdominal Visceral Fat Reduction in Obese Young Women. J Diabetes Res. 2017;2017:5071740. doi: 10.1155/2017/5071740. Epub 2017 Jan 1. PMID 28116314
- [Background] Cornelissen VA, Smart NA. Exercise training for blood pressure: a systematic review and meta-analysis. J Am Heart Assoc. 2013 Feb 1;2(1):e004473. doi: 10.1161/JAHA.112.004473. PMID 23525435
- [Background] Asmar R, Benetos A, Topouchian J, Laurent P, Pannier B, Brisac AM, Target R, Levy BI. Assessment of arterial distensibility by automatic pulse wave velocity measurement. Validation and clinical application studies. Hypertension. 1995 Sep;26(3):485-90. doi: 10.1161/01.hyp.26.3.485. PMID 7649586